CLINICAL TRIAL: NCT06126016
Title: A Multi-center, Prospective, Non-interventional, Observational Study to Evaluate the Efficacy and Safety of Pacitol Inj.(Paricalcitol) for Secondary Hyperparathyroidism With Stage 5D Chronic Kidney Disease (CKD 5D) Receiving Hemodialysis
Brief Title: A Observational Study to Evaluate the Efficacy and Safety of Pacitol Inj.
Status: Recruiting | Type: Observational
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BR-PCT-OS-401
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Chronic Kidney Disease 5D; Secondary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Secondary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of pacitol Inj.(paricalcitol) for secondary hyperparathyroidism with stage 5D chronic kidney disease (CKD 5D) receiving hemodialysis

ELIGIBILITY:
Inclusion Criteria:

* Among hemodialysis patients with secondary hyperparathyroidism due to chronic kidney disease (CKD 5D), those who are scheduled to administer Pacitol Inj. according to the product information.
* Those who voluntarily signed a written personal information collection and usage agreement to participate in this clinical study after receiving an explanation about the objective and methods of the study.
* Those able to understand this study, be cooperative in the execution of the study, and participate in the study until its completion.

Exclusion Criteria:

* Those with a history of hypersensitivity reactions to this drug or its components
* Those with evidence of vitamin D toxicity
* Those with hypercalcemia at enrollment
* Pregnant or lactating women
* Those with evidence of parathyroid adenoma who is scheduled to undergo parathyroidectomy.
* Those who have been administered with investigational drugs of other clinical trials within 12 weeks from the baseline(Visit 1).
* Those who are judged by the principle Investigator or sub-Investigator to be ineligible to participate in the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients with secondary hyperparathyroidism due to chronic kidney disease(CKD 5D)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects whose intact parathyroid hormone level applies to the therapeutic area(CKD 5D) | 12 weeks after administration

SECONDARY OUTCOMES:
Proportion of subjects whose intact parathyroid hormone level applies to the therapeutic area(CKD 5D) | 24 weeks after administration
Proportion of subjects whose intact parathyroid hormone level decreased by more than 30% | 12, 24 weeks compared to pre-dose
Incidence of anemia | From baseline to 12 weeks or 24 weeks
Change in intact parathyroid hormone | 12, 24 weeks compared to pre-dose
Change in Calcium X Phosphorus | 12, 24 weeks after administration

CONTACTS AND LOCATIONS:
Locations (1):
- DongGuk university Ilsan hospital, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No